CLINICAL TRIAL: NCT06085352
Title: An Investigator Initiated, Randomized, Single Center Clinical Study to Evaluate the Safety, Efficacy Using the TetraLens, a Tetracaine Releasing Therapeutic Bandage Contact Lens Undergoing a Photorefractive Keratotomy Procedure (PRK)
Brief Title: Evaluate the TetraLens, a Tetracaine Releasing Therapeutic Bandage Contact Lens in Patients Undergoing PRK Procedure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: USPFOS-01
Record Dates: First submitted 2023-09-26; First posted 2023-10-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Ocular Pain
Keywords: ocular pain
MeSH Terms: conditions — Eye Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Receive Investigational TetraLens BCL (Experimental): At random, one eye will receive the contact lens that contains the tetracaine HCL
  Interventions: Drug: TetraLens bandage contact lens
- Receive standard bandage contact lens (Sham Comparator): At random, one eye will receive the standard of care bandage contact lens
  Interventions: Device: Control Acuvue Oasys Bandage contact Lens

INTERVENTIONS:
Drug: TetraLens bandage contact lens — Methafilcon-A contact lens eluding tetracaine ophthalmic solution
  Arms: Receive Investigational TetraLens BCL
Device: Control Acuvue Oasys Bandage contact Lens — Standard of care bandage contact lens
  Arms: Receive standard bandage contact lens

SUMMARY:
The goal of this clinical trial is to determine the safety, efficacy, and comfort of the investigational TetraLens bandage contact lens in patients who have undergone photorefractive keratectomy (PRK). The main question[s] it aims to answer are:

* Understand benefit of managing pain following the surgical procedure
* Understand the safety of the Tetralens Participants will be asked to wear theTetraLens BCL in one eye for 6 days post-operatively and: document the daily quantity of oral analgesics needed and report ocular pain and contact lens comfort.

Researchers will compare the study lens in one eye to a control lens in the contralateral (other eye)

DETAILED DESCRIPTION:
The safety and efficacy of the methafilcon A and tetracaine HCL components of the TetraLens BCL have safety and efficacy profiles that are well established. This study aims to obtain the initial assessment of the safety efficacy and wearability of the TetraLens BCL for use a therapeutic bandage contact lens for short-term topical pain relief following ocular surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 22 years of age at time of surgery
2. patients who have been cleared to undergo PRK procedure
3. Patients who are willing to have procedure in both eyes, at least 1 week apart randomized to receive the product under investigation in one eye and control lens in other eye
4. Patients are able to wear bandage contact lens for 1 week
5. Patients able to attend all follow-up study visits

Exclusion Criteria:

1. Patients who have experienced complications during PRK procedures
2. Women of childbearing potential that are pregnant, nursing, or planning a pregnancy, and are not using effective methods of contraception. Effective contraception methods include:

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception. (Occasional abstinence is not an effective contraceptive method).
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least 6 weeks before Baseline. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
   3. Male sterilization (at least 6 months prior to Baseline). For female subjects in the study, the vasectomized male partner should be the sole partner for that subject
   4. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
   5. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
   6. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
3. Known allergy to Tetracaine or contraindications for its use
4. Significant anisometropia of greater than 2 diopters of manifest refraction spherical equivalent (MRSE) between eyes or hyperopes
5. Subjects having a history of previous eye surgery
6. Subjects with planned MRSE treatment of greater than 6.00D
7. Subjects with uncontrolled dry eye disease in the opinion of the investigator
8. History of systemic disorder such as diabetes, connective tissue disorder (systemic lupus erythematosis, rheumatoid arthritis, Sjögren syndrome, mucous membrane pemphigoid), thyroid disease, or immunosuppressive disorders (Human Immunodeficiency Virus [HIV], long-term steroid use, transplant recipient), that may affect post-operative healing
9. Corneal disease that may affect outcomes including keratoconus, form fruste keratoconus, limbal stem cell deficiency, pellucid marginal degeneration, contact lens warpage, and/or herpes keratitis
10. Use of chronic glaucoma and or hypotensive topical medications than in the view of the investigator could cause epitheliopathy and affect the rate of re-epithelization
11. Visually significant cataract
12. Other pathology of the cornea or anterior segment including lagophthalmos, blepharitis, anterior membrane dystrophy, corneal neuropathy, recurrent erosions and/or scarring that would affect wound re-epithelization
13. Use of medications that may affect and/or decrease the rate of corneal healing [e.g., systemic and or topical medications (corticosteroids, antimetabolites such as mitomycin) and/or antiviral medications] and or recent use (within the past 6 months) of isotretinoin, amiodarone or any medications that can affect corneal integrity
14. Any other factors that in the opinion of the investigator could put the subject at safety risk

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Efficacy of TetraLens BCL in the management of pain following surgical procedures | 6 days post-operative
  Cumulative number of daily pain medications up to Day 6 post-operative
Safety of TetraLens BCL | 6 days post-operative
  Corneal wound healing (re-epithelization)

CONTACTS AND LOCATIONS:
Overall Officials: Vance Thompson, MD, Principal Investigator — Vance Thompson Vision
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No